| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for A Phase I, Double-Blind,<br>Two-Part, Sequential Study to Evaluate the Pharmacokinetics<br>of Gepotidacin Tablets in Healthy Adult and Adolescent<br>Participants |
| <b>Compound Number</b> | : | GSK2140944 |
| <b>Effective Date</b> | : | 10-DEC-2019 |

# **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report (CSR) for Protocol GSK209611.
- This RAP is intended to describe the safety, tolerability, and pharmacokinetic (PK) analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) and Interim Analysis (IA) deliverable.

# **RAP Author(s):**

| PPD | | |
|---|---|---|
| Associate Bi<br>Services, PP | 10-DEC-2019 | |
| PPD Pharmacokin | eticist (Biostatistics, PPD) | 10-DEC-2019 |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Statistics Leader (Clinical Statistics) | 10-DEC-2019 | EMAIL |
| Programming Analyst (Clinical Programming) | 10-DEC-2019 | EMAIL |
| SM Executive Medical Director (Global Health Clinical) | 10-DEC-2019 | EMAIL |
| Clinical Development Director (R&D PCPS GCSD) | 10-DEC-2019 | EMAIL |
| Manager (Clinical Data Management) | 10-DEC-2019 | EMAIL |
| Director (CPMS) | 10-DEC-2019 | EMAIL |
| Medical Director SERM (SMG Pharma Safety) | 10-DEC-2019 | EMAIL |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval<br>Method |
|---------------------------------|-------------|--------------------|
| Director (Clinical Statistics) | 10-DEC-2019 | EMAIL |
| Director (Clinical Programming) | 10-DEC-2019 | EMAIL |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | DDUCTIO | N | 5 |
| 2. | SUMN | ARY OF | KEY PROTOCOL INFORMATION | 5 |
| ۷. | 2.1. | | s to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | • | bjective(s) and Endpoint(s) | |
| | 2.3. | | esign | |
| | 2.4. | | al Analyses | |
| | 2. 1. | Otationo | ai / tilaiy 000 | |
| 3. | PLAN | NED ANA | LYSES | 9 |
| | 3.1. | | Analyses | |
| | 3.2. | | alyses | |
| 4 | ANIAL | Vele Doi | ZULI ATIONIC | 40 |
| 4. | 4.1. | | PULATIONS | |
| | 4.1. | Protocol | Deviations | 10 |
| 5. | CONS | SIDERATI | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | ENTIONS | S | 11 |
| | 5.1. | | e Definitions | 11 |
| | 5.2. | | onsiderations for Data Analyses and Data Handling | |
| | | Convent | tions | 11 |
| _ | | | | |
| 6. | | | ATION ANALYSES | |
| | 6.1. | Overvie | w of Planned Study Population Analyses | 13 |
| 7. | DLAD | MACOKII | NETIC ANALYSES | 1.1 |
| ١. | 7.1. | | Pharmacokinetic Analyses | |
| | 7.1. | 7.1.1. | Endpoint / Variables | |
| | | 7.1.1. | 7.1.1.1. Drug Concentration Measures | |
| | | | 7.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 7.1.2. | Summary Measure | |
| | | 7.1.3. | Population of Interest | |
| | | 7.1.4. | Statistical Analyses / Methods | |
| | | | 7.1.4.1. Statistical Methodology Specification | |
| | 7.2. | Seconda | ary Pharmacokinetic Analyses | |
| | | 7.2.1. | Endpoint / Variables | |
| | | | 7.2.1.1. Derived Pharmacokinetic Parameters | 16 |
| | | 7.2.2. | Summary Measure | 16 |
| | | 7.2.3. | Population of Interest | 17 |
| | | 7.2.4. | Statistical Analyses / Methods | 17 |
| | | | 7.2.4.1. Statistical Methodology Specification | 17 |
| _ | 0455 | T\/ | V050 | 40 |
| 8. | | | YSES | |
| | 8.1.<br>8.2. | | Events Analyses | |
| | 0.2. | 8.2.1. | Events of Special Interest Analyses | |
| | 8.3. | - | Acetylcholinesterase-Inhibition AESIsLaboratory Analyses | |
| | 8.4. | | afety Analyses | |
| | ∪. <del>-</del> †. | Ouilei O | aloty / thatysos | 20 |
| 0 | DEEE | DENCES | | 24 |

| ١0. | APPE | NDICES | | 22 |
|---|---|---|---|---|
| | 10.1. | Appendix | 1: Schedule of Activities | 22 |
| | | 10.1.1. | Protocol Defined Time and Events Table | 22 |
| | | 10.1.2. | Protocol Defined Safety and PK Assessments | 27 |
| | 10.2. | | 2: Study Phases and Treatment Emergent Adverse | |
| | | Events | | 31 |
| | | 10.2.1. | Treatment States | |
| | | | 10.2.1.1. Treatment States for Safety Data | 31 |
| | | | 10.2.1.2. Treatment States for AE Data | |
| | | | 10.2.1.3. Study Phases for Concomitant Medication | |
| | | 10.2.2. | Treatment Emergent Flag for Adverse Events | |
| | 10.3. | | 3: Data Display Standards & Handling Conventions | |
| | | 10.3.1. | Study Treatment & Sub-group Display Descriptors | |
| | | 10.3.2. | Reporting Process & Standards | 33 |
| | | 10.3.3. | Reporting Standards for Pharmacokinetics | 35 |
| | 10.4. | | 4: Derived and Transformed Data | |
| | | 10.4.1. | General | |
| | | 10.4.2. | Study Population | |
| | | 10.4.3. | Safety | |
| | 10.5. | | 5: Reporting Standards for Missing Data | |
| | | 10.5.1. | Premature Withdrawals | |
| | | 10.5.2. | Handling of Missing Data | |
| | | | 10.5.2.1. Handling of Missing and Partial Dates | |
| | 10.6. | | 6: Values of Potential Clinical Importance | |
| | | | ECG | |
| | | | Vital Signs | 39 |
| | 10.7. | Appendix | 7: Division of Microbiology and Infectious Diseases Adult | |
| | | | Tables for Adverse Events Assessments (2007) | |
| | 40.0 | | Laboratory Values | |
| | 10.8. | | 8: Multiple Comparisons & Multiplicity | |
| | | 10.8.1. | Handling of Multiple Comparisons & Multiplicity | |
| | 10.9. | | s 9: Abbreviations & Trade Marks | |
| | | | Abbreviations | |
| | 40.40 | | Trademarks | |
| | 10.10. | | 10: List of Data Displays | |
| | | | Data Display Numbering | |
| | | | Mock Example Shell Referencing | |
| | | | Deliverables | |
| | | | Study Population Tables | |
| | | | Safety Tables | |
| | | | Safety Figures | |
| | | | Pharmacokinetic Tables | |
| | | | Pharmacokinetic Figures | |
| | | | ICH Listings | |
| | | 10.10.10 | Non-ICH Listings | 58 |

### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the CSR for Protocol GSK209611

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes to the planned statistical analysis specified in the protocol (Dated: 13-JUN-2019) are listed below.

- For adolescent serum creatinine lab data, pediatric DMID toxicity criteria will be used.
- Events associated with acetylcholinesterase inhibition will be programmatically and manually assessed as adverse events of special interest (AESIs). See analysis plan in Section 8.2 and Section 10.4.3.
- Section 7.1.1.2 of this analysis plan specifies that the accumulation ratio Ro AUC will be calculated as AUC( $0-\tau$ ) after the second dose divided by AUC( $0-\tau$ ) after the first dose (rather than using AUC(0-6) as stated in the protocol), to make this formula widely applicable to all dosing intervals.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate the pharmacokinetics (PK) of a single 1500- milligrams (mg) dose and two 3000-mg doses of gepotidacin given 6 and 12 hours apart in adult participants | <ul> <li>1500 mg single dose</li> <li>Plasma gepotidacin AUC(0-t), AUC(0-∞), AUC(0-24), AUC(0-48), and Cmax, as data permit</li> <li>3000 mg two doses</li> <li>Plasma gepotidacin AUC(0-t), AUC(0-т), AUC(0-24), AUC(0-48), Ro (accumulation ratio), and Cmax, as data permit</li> </ul> |

#### 209611

# Part 2

 To evaluate the PK of a single 1500-mg dose and two 3000-mg doses of gepotidacin given at a dosing interval (to be determined) in adolescent participants

#### 1500 mg single dose

 Plasma gepotidacin AUC(0-t), AUC(0-∞), AUC(0-24), AUC(0-48), and Cmax, as data permit

## 3000 mg two doses

 Plasma gepotidacin AUC(0-t), AUC(0-τ), AUC(0-24), AUC(0-48), Ro (accumulation ratio), and Cmax, as data permit

#### Parts 1 and 2

 To assess the safety of gepotidacin in adult participants and adolescent participants  Adverse events, clinical laboratory tests, vital signs (systolic and diastolic blood pressure and heart rate), and 12-lead electrocardiogram readings

#### Secondary

#### Part 1

 To assess the urine PK of gepotidacin following a single 1500-mg dose and two 3000-mg doses of gepotidacin given 6 and 12 hours apart in adult participants  Urine endpoints include Ae total, Ae(t1-t2), AUC(0-t), AUC(0-24), AUC(0-48), percentage of the given dose of drug excreted in urine (fe%), and renal clearance of drug (CLr) of gepotidacin, as data permit

#### Part 2

 To assess the urine PK of gepotidacin following a single 1500-mg dose and two 3000-mg doses of gepotidacin given at a dosing interval (to be determined) in adolescent participants  Urine endpoints include Ae total, Ae(t1-t2), AUC(0-τ), AUC(0-24), AUC(0-48), fe%, and CLr of gepotidacin, as data permit

#### Parts 1 and 2

To assess the plasma PK of gepotidacin

 Plasma gepotidacin Tmax, tlag, and t1/2, as data permit

# 2.3. Study Design



Note: Participants will be randomized in in a 14:3 ratio in order to obtain 12 evaluable participants on active treatment and 2 evaluable participants on placebo.

# Design Features

- Phase I, double-blind, single-center, randomized, sequential, two-part study
- Part 1: Participants will be randomly assigned to receive either all active treatment (gepotidacin) or placebo for all 3 periods. Approximately 17 participants will be randomized (in a 14:3 ratio) to receive a single dose of gepotidacin 1500 mg (Treatment A) or matching placebo (Treatment B) in Period 1, gepotidacin 3000 mg separated by 12 hours (Treatment C) or matching placebo (Treatment D) in Period 2, and gepotidacin 3000 mg separated by 6 hours (Treatment E) or matching placebo (Treatment F) in Period 3 to obtain 12 evaluable participants on active treatment and 2 evaluable participants on placebo.
- Part 2: Participants will be randomly assigned to receive either all active treatment (gepotidacin) or placebo for both periods. Approximately 17 participants will be randomized (in a 14:3 ratio) to receive a single dose of gepotidacin 1500 mg (Treatment A) or matching placebo (Treatment B) in Period 1, and gepotidacin 3000 mg (Treatment G) or matching placebo (Treatment H) in Period 2 to obtain 12 evaluable participants on active treatment and 2 evaluable participants on placebo.
- In Part 2, the interval for the two 3000-mg doses in Period 2 will be between 6 hours and 12 hours based on the PK and safety results from Part 1.

# The GlaxoSmithKline group of companies

| Dosing | Part 1 – Adult Participants: |
|---|---|
| | Treatment A: Single dose 1500 mg (Period 1) |
| | Treatment B: Matching placebo (Period 1) |
| | Treatment C: Two 3000 mg doses given at Hour 0 and Hour 12 (Period 2) |
| | Treatment D: Two matching placebo doses given at Hour 0 and Hour 12 (Period 2) |
| | Treatment E: Two 3000 mg doses given at Hour 0 and Hour 6 (Period 3) |
| | <ul> <li>Treatment F: Two matching placebo doses given at Hour 0 and Hour 6<br/>(Period 3)</li> </ul> |
| | Part 2 - Adolescent Participants |
| | Treatment A: Single dose 1500 mg (Period 1) |
| | Treatment B: Matching placebo (Period 1) |
| | Treatment G: Two 3000 mg doses (Period 2; exact dosing interval to be determined after Part 1 is complete) |
| | Treatment H: Two matching placebo doses (Period 2; exact dosing interval to be determined after Part 1 is complete) |
| Time and Events | See Appendix 1: Schedule of Activities (SoA) |
| Treatment<br>Assignment | Part 1 – Adult Participants: Participants will be randomly assigned to receive either all active treatment (gepotidacin, Treatment A/C/E) or placebo (Treatment B/D/F) for all 3 periods |
| | Part 2 – Adolescent Participants: Participants will be randomly assigned to receive either all active treatment (gepotidacin, Treatment A/G) or placebo (Treatment B/H) for both periods. |
| Interim<br>Analysis | The interim analysis will consist data management listings and WinNonLin outputs. Preliminary plasma PK and safety results from participants in Part 1 will be reviewed by the sponsor before enrolling participants into the next part of the study. The dosing interval to be used when two gepotidacin doses are given in Part 2, Period 2 will be determined after a review of the PK and safety results from Part 1. The number of PK samples and the PK sampling time points may be modified based on the adult PK data from Part 1. |
| | An ad hoc review of 12-lead electrocardiogram (ECG) data may be performed between Part 1, Period 2 and Part 1, Period 3. |

# 2.4. Statistical Analyses

There is no formal research hypothesis that will be statistically tested in this study.

### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

The interim analysis will consist data management listings and WinNonLin outputs. Preliminary plasma PK and safety results from participants in Part 1 will be reviewed by the sponsor before enrolling participants into the next part of the study. The dosing interval to be used when two gepotidacin doses are given in Part 2, Period 2 will be determined after a review of the PK and safety results from Part 1. The number of PK samples and the PK sampling time points may be modified based on the adult PK data from Part 1.

An ad hoc review of 12-lead ECG data may be performed between Part 1, Period 2 and Part 1, Period 3.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Enrolled | All participants who sign the ICF/assent. | Study Population |
| Randomized | All participants who are randomized. | Study Population |
| Safety | All participants who take at least 1 dose of study intervention. | <ul><li>Study Population</li><li>Safety</li></ul> |
| PK | Participants who receive at least 1 dose of gepotidacin and have evaluable postdose plasma concentration data for gepotidacin. | PK Concentration |
| PK Parameter | All participants in the PK population who | PK parameter |
| | received gepotidacin for whom valid and evaluable plasma PK parameters are derived for gepotidacin. | PK statistical analysis |

#### NOTES:

 Please refer to Appendix 10: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorized on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

### 5.1. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the last available assessment prior to time of study drug administration, unless noted otherwise.

| Parameter | Study Assessments Considered as Baseline | | | | Baseline |
|---|---|---|---|---|---|
| | Screening | Day -<br>1 | Day 1 (Pre-<br>Dose) for Part<br>1 Period 1 and<br>Part 2 all<br>Periods | Day 5 (Pre-Dose)<br>and Day 9 (Pre-<br>Dose) for Part 1<br>Period 2 and 3 | Used in Data<br>Display |
| | Safety | | | | |
| Hematology | Х | Х | | | Day -1 |
| Chemistry | Х | Х | | | Day -1 |
| Routine<br>Urinalysis | X | Х | | | Day -1 |
| 12-Lead ECG | X | Х | Х | Х | Day 1, Day 5<br>and Day 9<br>Pre-Dose |
| Vital Signs | Х | Х | Х | Х | Day 1, Day 5<br>and Day 9<br>Pre-Dose |

**NOTES:** unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

If baseline data of ECG or Vital Signs is missing, substitute missing data with the Day -1 or the last non-missing baseline value, whichever date/time is closer to the reference date/time.

For any other assessment, if baseline data is missing no derivation will be performed and baseline will be set to missing, unless otherwise stated.

# 5.2. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

# The GlaxoSmithKline group of companies

| Section | Component |
|---------|----------------------------------------------------------------|
| 10.1 | Appendix 1: Schedule of Activities |
| 10.2 | Appendix 2: Study Phases and Treatment Emergent Adverse Events |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Reporting Standards for Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.7 | Appendix 7: Division of Microbiology and Infectious Disease |
| 10.8 | Appendix 8: Multiple Comparisons and Multiplicity |
| 10.9 | Appendix 9: Abbreviations & Trade Marks |
| 10.10 | Appendix 10: List of Data Displays |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Enrolled, Randomized, and Safety population, unless otherwise specified.

Study population analyses including analyses of subjects enrolled by Country and Site ID, subject's disposition, screening failures, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 10: List of Data Displays.

# 7. PHARMACOKINETIC ANALYSES

# 7.1. Primary Pharmacokinetic Analyses

# 7.1.1. Endpoint / Variables

#### 7.1.1.1. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Standards for Pharmacokinetic). Only total gepotidacin plasma PK concentrations will be measured and reported in the bioanalytical data. Therefore, unbound plasma PK concentrations will be derived by multiplying the total plasma PK concentrations by 0.67, to correct for the low plasma protein binding of gepotidacin (33%) observed in previous studies.

#### 7.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (8.0 or higher). All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permit.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the plasma concentration-time curve from time 0 (predose) to the last |
| | quantifiable concentration, to be calculated using the linear trapezoidal rule for each |
| | incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-∞) | Area under the concentration-time curve from time 0 (predose) extrapolated to infinite time, |
| | to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log |
| | trapezoidal rule for each decremental trapezoid. (Calculated for single dose administration) |
| AUC(0-24) | Area under the plasma concentration-time curve from time 0 (predose) to the concentration |
| | at 24 hours postdose (post first dose for periods where 2 doses are administered), to be |
| | calculated using the linear trapezoidal rule for each incremental trapezoid and the log |
| | trapezoidal rule for each decremental trapezoid. |
| AUC(0-48) | Area under the plasma concentration-time curve from time 0 (predose) to the concentration |
| | at 48 hours postdose (post first dose for periods where 2 doses are administered), to be |
| | calculated using the linear trapezoidal rule for each incremental trapezoid and the log |
| | trapezoidal rule for each decremental trapezoid. |
| $AUC(0-\tau)$ | Area under the concentration-time curve from time 0 (predose) to time tau (tau = 12 and 6 |
| | for Part 1, Periods 2 and 3, respectively; for Part 2, tau will be between 6 and 12) |
| | (Calculated for periods where 2 doses are administered) |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Ro AUC | Accumulation ratio calculated as AUC(0-т) after the second dose, where 0 is the timepoint |
| | prior to second dose, divided by AUC(0-τ) after the first dose, where 0 is the predose |
| | timepoint prior to the first dose. (Calculated for periods where 2 doses are administered) |
| Ro Cmax | Accumulation ratio calculated as Cmax after the second dose divided by Cmax after the first |
| | dose. (Calculated for periods where 2 doses are administered) |

## NOTES:

Additional parameters may be included as required.

## 7.1.2. Summary Measure

#### Part 1

Pharmacokinetic parameters AUC(0-t),  $AUC(0-\infty)$  (Period 1), AUC(0-24), AUC(0-48),  $AUC(0-\tau)$  (Part 1 Periods 2 and 3), Cmax, RO AUC (Part 1 Period 2 and 3), and RO Cmax (Part 1 Period 2 and 3) following a single 1500 mg dose of gepotidacin (Part 1 Period 1) and two 3000 mg doses of gepotidacin (Part 1 Periods 2 and 3) in healthy adult participants will be summarized by treatment. Gepotidacin PK parameter estimates will be listed by participant and treatment.

#### Part 2

Pharmacokinetic parameters AUC(0-t), AUC(0-∞) (Part 2 Period 1), AUC(0-24), AUC(0-48), AUC(0-τ) (Part 2 Period 2), Cmax, RO AUC (Part 2 Period 2), and RO Cmax (Part 2 Period 2) following a single 1500 mg dose of gepotidacin (Part 2 Period 1) and two 3000 mg doses of gepotidacin at a time interval determined based on data from Part 1 (Part 2 Period 2) in healthy adolescent participants will be summarized by treatment. Gepotidacin PK parameter estimates will be listed by participant and treatment.

#### 7.1.3. Population of Interest

The primary PK analyses will be based on the PK population for plasma PK concentrations and the PK parameter population for plasma PK parameters.

# 7.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Section 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/ variables defined in Section 7.1.1 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed.

Primary plasma PK parameters AUC(0-t), AUC(0-∞) (Period 1), AUC(0-24), AUC(0-48), AUC(0-τ) (Periods 2 and 3), Cmax, RO AUC (Periods 2 and 3), and RO Cmax (Periods 2 and 3) will be estimated for gepotidacin. For each of these parameters the following summary statistics will be calculated by Study Part and treatment: median, maximum, minimum, arithmetic mean, SD, 95% confidence interval (CI) for the arithmetic mean, geometric mean, CV on geometric mean, 95% CI for the geometric mean, and SD of logarithmically transformed data.

#### 7.1.4.1. Statistical Methodology Specification

There are no planned statistical PK analyses additional to summary statistics.

# 7.2. Secondary Pharmacokinetic Analyses

# 7.2.1. Endpoint / Variables

#### 7.2.1.1. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin (8.0 or higher) or using the currently supported version of SAS (9.4 or higher). All calculations of non-compartmental parameters will be based on actual sampling times.

Plasma/urine pharmacokinetic parameters listed below will be determined from the plasma/urine concentration-time data, as data permit.

| Parameter | Parameter Description |
|---|---|
| Ae total | Total unchanged drug (total amount of drug excreted in urine), calculated by adding |
| | all the fractions of drug collected over all the allotted time intervals |
| Ae(t1-t2) | Amount of drug excreted in urine in time intervals of predose, 0 to 2 hours, 2 to 4 |
| | hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, 36 to |
| | 48 hours, and 48 to 60 hours (Part 1, Period 2 and Period 3) after dosing |
| AUC(0-т) | Area under the concentration-time curve from time 0 (predose) to time tau (tau = 12 |
| | and 6 for Part 1, Periods 2 and 3, respectively; for Part 2, tau will be between 6 and |
| | 12) (urine) |
| AUC(0-24) | Area under the concentration-time curve from time 0 (predose) to 24 hours postdose |
| | administration following the first dose (urine) |
| AUC(0-48) | Area under the concentration-time curve from time 0 (predose) to 48 hours postdose |
| | administration following the first dose (urine) |
| fe% | Percentage of the given dose of drug excreted in urine, calculated as: |
| | fe% = (Ae total/Dose) × 100% |
| CLr | Renal clearance of drug, calculated as: Ae total/AUC(0-t) |
| Tmax | Time to reach maximum observed plasma concentration |
| tlag | Lag time before observation of drug concentrations in plasma |
| t1/2 | Apparent terminal phase half-life (plasma) |

#### NOTES:

Additional parameters may be included as required.

# 7.2.2. Summary Measure

#### Part 1

Urine PK parameters Ae total, Ae(t1-t2), AUC(0-τ) (Periods 2 and 3), AUC(0-24), AUC(0-48), fe%, and CLr, and plasma PK parameters Tmax, Tlag, and t1/2 following a single 1500 mg dose of gepotidacin (Part 1 Period 1) and two 3000 mg doses of gepotidacin (Part 1 Periods 2 and 3) in healthy adult participants will be summarized by treatment. Gepotidacin PK parameter estimates will be listed by participant and treatment.

Part 2

Urine PK parameters Ae total, Ae(t1-t2), AUC(0-τ) (Period 2), AUC(0-24), AUC(0-48), fe%, and CLr and plasma PK parameters Tmax, Tlag, and t1/2 following a single 1500 mg dose of gepotidacin (Part 2 Period 1) and two 3000 mg doses of gepotidacin at a time interval to be determined from Part 1 (Part 2 Period 2) in healthy adolescent participants will be summarized by treatment. Gepotidacin PK parameter estimates will be listed by participant and treatment.

## 7.2.3. Population of Interest

The secondary PK analyses will be based on the PK population for urine/plasma PK concentrations, and the PK parameter population for urine/plasma PK parameters.

# 7.2.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 7.2 will be summarized using descriptive statistics, graphically presented (where appropriate) and listed.

Secondary urine PK parameters Ae total, Ae(t1-t2), AUC(0-τ), AUC(0-24), AUC(0-48), fe%, and CLr, and plasma PK parameters Tmax, Tlag, and t1/2 will be estimated for gepotidacin. For each of these parameters the following summary statistics will be calculated by Study Part and treatment: median, maximum, minimum, arithmetic mean, SD, 95% CI for the arithmetic mean, geometric mean, CV on geometric mean, 95% CI for the geometric mean, and SD of logarithmically transformed data.

# 7.2.4.1. Statistical Methodology Specification

There are no planned statistical PK analyses additional to summary statistics.

### 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

# 8.1. Adverse Events Analyses

The severity of AEs and SAEs will be determined by the investigator according to the US National Institute of Allergy and Infectious Diseases Division of Microbiology and Infectious Diseases (DMID) criteria for adult toxicity assessment, with the exception of serum creatinine adolescent laboratory data, which will be assessed using pediatric toxicity criteria. All reported AEs will be coded using MedDRA and summarized by system organ class (SOC) and preferred term (PT).

Adverse event severity is classified as mild (grade = 1), moderate (grade = 2), severe (grade = 3), potentially life threatening (grade = 4) or resulting in death (grade = 5). Adverse events starting after the first dose of study treatment with a missing severity will be classified as severe. If a participant reports an AE more than once within an SOC/PT, the AE with the worst-case severity will be used in the corresponding severity summaries.

Relationship to study treatment, as indicated by the investigator, is classified as "not related" or "related". Adverse events with a missing relationship to study treatment will be regarded as "related" to study treatment. If a participant reports the same AE more than once within an SOC/PT, the AE with the worst-case relationship to study treatment will be used in the corresponding relationship summaries.

Adverse events analyses including the analysis of AEs, SAEs and other significant AEs will be based on GSK Core Data Standards. All AEs, study drug related AEs, SAEs, and AEs leading to discontinuation of study treatment or withdrawal from study will be provided in separate listings. The relationship between SOC and PT will be listed. Summary tables will be provided by SOC, PT, and maximum grade.

In summary tables where AEs are presented by SOC, PT, and maximum grade, SOCs will be sorted in descending order of the total incidence then alphabetically, PTs will be sorted in descending order of the total incidence then alphabetically within the SOC.

For completely missing or partial missing AE start date or end date, imputation rules will be applied following Section 10.4.1.

In addition, a summary of the number and percentage of participants with common AEs, defined as AEs with  $\geq$ 5% incidence in any treatment group, will be presented in descending order of total incidence by PT. The details of the planned displays are provided in Appendix 10: List of Data Displays.

# 8.2. Adverse Events of Special Interest Analyses

Cardiovascular, Gastrointestinal Adverse Events and events related to Acetylcholinesterase inhibition as determined by algorithm will be considered AEs of Special Interest (AESIs). AESIs except those for Acetylcholinesterase inhibition, are flagged in the eCRF and details of events are collected on special eCRF pages. Acetylcholinesterase-Inhibition AESIs will be programmatically matched with the list of AEs specified in Section 8.2.1. In addition, there will be a manual review of AE listings to ensure accuracy and completeness of AESI reporting.

# 8.2.1. Acetylcholinesterase-Inhibition AESIs

Any reported AE listed in the table below with a start time no later than 12 hours after the last dose administered in each treatment period, as evaluated by the investigator as per the DMID grading criteria provided in protocol Section 10.8 Appendix 8: Division of Microbiology and Infectious Disease Adult Toxicity Tables for Adverse Event Assessment, will be programmatically identified as Acetylcholinesterase inhibition related AESI.

Table 1 List of AEs for programming to be considered due to Acetylcholinesterase-Inhibition

- Respiratory
  - Bronchospasm (acute)
  - o Dyspnea
  - o Bronchorrhea
- Gastrointestinal
  - o Nausea
  - o Vomiting
  - o Diarrhea
  - o GI cramping and pain
- Cardiovascular
  - o Bradycardia
- Neurological
  - Seizure/Convulsions
  - Vasovagal syncope
  - Salivation
  - Lacrimation
  - Diaphoresis/sweating

AESIs will be listed and tabulated, and a Cumulative Grade will be determined, calculated by the sum of the grade of each reported AE. This enables both the number of AEs and the severity of each AE to be taken into account. For instance, if two AEs in the table above are reported, one of Grade 1 and the other of Grade 3 according to DMID, the total grade of 4 would result in a Cumulative Grade 2 per Table 2 below.

Table 2 Cumulative Grading of Acetylcholinesterase AESI

| | Cumulative | Cumulative | Cumulative | Cumulative |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Total Grade of<br>Signs & Symptoms | 1 to 3 | 4 to 6 | 7 to 10 | ≥ 11 |

The details of the planned displays are provided in Appendix 10: List of Data Displays.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of chemistry laboratory tests, hematology laboratory tests, urinalysis, and liver function tests will be based on GSK Core Data Standards. Division of Microbiology and Infectious Diseases (DMID) grading for all parameters as specified in the protocol will be assigned programmatically by PPD in the Laboratory Analysis Dataset. The details of the planned displays are in Appendix 10: List of Data Displays.

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 10: List of Data Displays.

# 9. REFERENCES

GlaxoSmithKline Document Numbers 2019N401436\_00 (Original – 04-JUN-2019): A Phase I, Double-Blind, Two-Part, Sequential Study to Evaluate the Pharmacokinetics of Gepotidacin Tablets in Healthy Adult and Adolescent Participants (04-JUN-2019).

# 10. APPENDICES

# 10.1. Appendix 1: Schedule of Activities

# 10.1.1. Protocol Defined Time and Events Table

Table 3 Part 1 Adult Participants

| Procedure <sup>1</sup> | Check<br>-in | | | at Period 1<br>ays) | | | | t Period 2<br>ays) | | Trea | atment Per<br>(Days) | riod 3 | Follow-up (7 [±3] days after last dose) or Early Termination | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | | |
| Confined to clinic | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Inclusion and exclusion criteria | Х | | | | | | | | | | | | | Recheck clinical<br>status before<br>study<br>intervention |
| Brief physical examination <sup>2</sup> | Х | | | | | | | | | | | Х | Х | |
| Pregnancy test | х | | | | | | | | | | | | Х | Urine pregnancy<br>test (if WOCBP),<br>as appropriate<br>(see Table 10 in<br>Protocol) |
| Drug, alcohol, and cotinine screen | Х | | | | | | | | | | | | | See Table 10 in<br>Protocol |

2019N422403\_00

209611

| Procedure <sup>1</sup> | Check<br>-in | | Treatmen<br>(Da | | | | | t Period 2<br>lys) | | Trea | tment Per<br>(Days) | iod 3 | Follow-up<br>(7 [±3] days<br>after last<br>dose) or<br>Early<br>Termination | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | | |
| Laboratory assessments | х | | | | Х | | | | Х | | | Х | х | Including serum<br>chemistry,<br>hematology, and<br>urinalysis (see<br>Appendix 2 in<br>Protocol) |
| 12-lead ECG <sup>3</sup> | Х | X | X | X | | X | X | Х | | X | Х | Х | х | See Table 4,<br>Table 5, and<br>Table 6 for<br>timing of<br>assessments |
| ECG Holter<br>monitoring <sup>4</sup> | Х | X | Х | | Х | Х | Х | | Х | Х | Х | | | See Table 4,<br>Table 5, and<br>Table 6 for<br>timing of<br>assessments |
| Vital signs | Х | Х | Х | Х | | Х | Х | Х | | Х | Х | Х | Х | See Table 4,<br>Table 5, and<br>Table 6 for<br>timing of<br>assessments |
| Study intervention | | Х | | | | Х | | | | Х | | | | See Table 4,<br>Table 5, and<br>Table 6 for time<br>points |

# 2019N422403 00

209611

| Procedure <sup>1</sup> | Check<br>-in | | | t Period 1<br>lys) | | | Treatmen<br>(Da | t Period 2<br>ys) | | Trea | tment Per<br>(Days) | iod 3 | Follow-up<br>(7 [±3] days<br>after last<br>dose) or<br>Early<br>Termination | Notes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <b>-1</b> | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | | |
| Blood collection for pharmacokinetics | | Х | | | | Х | Х | Х | | Х | Х | Х | | See Table 4,<br>Table 5, and<br>Table 6 for time<br>points |
| Urine collection for pharmacokinetics | | Х | Х | Х | | Х | Х | Х | | Х | Х | х | | See Table 4,<br>Table 5, and<br>Table 6 for time<br>points |
| AE/SAE review | Х | <b>←====</b> | | ====== | ====== | | | | | | ====== | :====> | Х | |
| Concomitant medication review | Х | <b>←====</b> | ====== | ====== | ====== | ====== | ====== | | ====== | | | ·====> | Х | |

AE = adverse event, ECG = electrocardiogram, SAE = serious AE; WOCBP = woman of childbearing potential.

- When coinciding with safety and/or pharmacokinetic assessments, ECGs, vital signs, and pharmacokinetic blood collections should be performed in said order.
- A brief physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).
- Triplicate 12-lead ECGs will be measured on Day -1.
- ECG Holter monitoring will begin approximately 12 hours prior to first dose until 24 hours after dosing of each treatment period.

209611

**Table 3: Part 2 Adolescent Participants** 

| Dra and wat | Check-in | Tre | atment Perio | od 1 | Check-<br>in <sup>2</sup> | Tre | eatment Perio | od 2 | Follow-up<br>(7 [±3] days | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure <sup>1</sup> | -1 | 1 | 2 | 3 | -1 | 1 | 2 | 3 | after last<br>dose) or Early<br>Termination | Notes |
| Confined to clinic | Х | X | Х | Х | Х | Х | Х | X | | Treatment Period 1 and<br>Treatment Period 2 may be<br>separated by 7 days but no<br>more than 10 days. |
| Inclusion and exclusion criteria | Х | | | | Х | | | | | Recheck clinical status before study intervention |
| Brief physical examination <sup>3</sup> | Χ | | | | Х | | | Х | X | |
| Pregnancy test | Х | | | | X | | | | Х | Urine pregnancy test (if WOCBP), as appropriate (see Table 10 in Protocol) |
| Drug, alcohol, and cotinine screen | Х | | | | Х | | | | | See Table 10 in Protocol |
| Laboratory assessments | Х | | | X | Х | | | Х | Х | Including serum chemistry,<br>hematology, and urinalysis<br>(see Appendix 2 in<br>Protocol) |
| 12-lead ECG <sup>4</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | See Table 7, Table 8, and<br>Table 9 for timing of<br>assessments |
| ECG Holter monitoring <sup>5</sup> | X | Χ | X | | X | X | Х | | | See Table 7, Table 8, and Table 9 for timing of assessments |
| Vital signs | X | Χ | Х | Х | Х | X | Х | Х | Х | See Table 7, Table 8, and Table 9 for timing of assessments |
| Study intervention | | Χ | | | | Х | | | | See Table 7, Table 8, and Table 9 for time points |

# 2019N422403 00

209611

| Procedure <sup>1</sup> | Check-in | Tre | eatment Perio | od 1 | Check-<br>in <sup>2</sup> | Tre | atment Perio | od 2 | Follow-up<br>(7 [±3] days<br>after last | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Frocedure | -1 | 1 | 2 | 3 | -1 | 1 | 2 | 3 | dose) or Early Termination | Notes |
| Blood collection for pharmacokinetics | | Х | Х | Х | | Х | Х | Х | | See Table 7, Table 8, and Table 9 for time points |
| Urine collection for pharmacokinetics | | Х | Х | Х | | Х | Х | Х | | See Table 7, Table 8, and Table 9 for time points |
| AE/SAE review | Х | <b>←====</b> | ======= | | | | | ====== | Х | |
| Concomitant medication review | Х | <b>←====</b> | ======= | ======= | ======= | | | =====> | Х | |

AE = adverse event, ECG = electrocardiogram, SAE = serious AE; WOCBP = woman of childbearing potential.

- When coinciding with safety and/or pharmacokinetic assessments, ECGs, vital signs, and pharmacokinetic blood collections should be performed in said order.
- <sup>2</sup> Check-in procedures only necessary if participant leaves the clinic between Treatment Period 1 and Treatment Period 2.
- A brief physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).
- <sup>4</sup> Triplicate 12-lead ECGs will be measured on Day -1 (before each treatment period).
- <sup>5</sup> ECG Holter monitoring will begin approximately 12 hours prior to first dose until 24 hours after dosing of each treatment period.

# 10.1.2. Protocol Defined Safety and PK Assessments

Table 4 Safety and PK Assessments - Part 1, Period 1

| Procedure <sup>1</sup> | | | | | | | | | t Period '<br>nt (hours | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Predose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 6 | 8 | 12 | 24 | 36 | 48 |
| 12-lead ECG <sup>2</sup> | Х | | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | Х |
| ECG Holter monitoring | Х | | X | | | | | | | | | | | | |
| Vital signs | Х | | | | Х | Х | | | Х | | Х | Х | Х | Χ | Х |
| Study intervention | | Х | | | | | | | | | | | | | |
| Blood PK sample | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х |
| Urine PK collection <sup>3</sup> | Х | | ) | X | | | Х | | Х | Х | Х | Х | Х | Χ | Х |

ECG = electrocardiogram; PK = pharmacokinetic.

- When coinciding with safety and/or PK assessments, ECGs, vital signs, and PK blood collections should be performed in said order.
- Triplicate 12-lead ECGs will be measured at predose. Single 12-lead ECGs will be measured at all other time points.
- Urine collection intervals include 0 (predose), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours.

Table 5 Safety and PK Assessments - Part 1, Period 2 (12-Hour Dose Interval)

| | | | | | | | | | | | atmen | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure <sup>1</sup> | | | | | | | | | | Tim | e poi | nt (ho | urs) | | | | | | | | | | | | |
| | Predose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 6 | 8 | 12 | 12.5 | 13 | 13.5 | 14 | 14.5 | 15 | 16 | 18 | 20 | 24 | 36 | 48 | 60 |
| 12-lead ECG <sup>2</sup> | Х | | Х | Χ | Х | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х |
| ECG Holter monitoring | Х | | | | | | | | | | Χ | | | | | | | | | | | | | | |
| Vital signs | Χ | | | | Χ | Χ | | | Χ | | Χ | Χ | | | Χ | Χ | | | | Χ | | Χ | Χ | Χ | Χ |
| Study intervention | | Χ | | | | | | | | | | Х | | | | | | | | | | | | | |
| Blood PK sample | Х | | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Χ | Х | Х | Х |
| Urine PK collection <sup>3</sup> | Х | | Х | | | | Х | | Х | Χ | Х | | | X | | | Х | • | Х | Х | Х | Χ | Х | Х | Х |

ECG = electrocardiogram; PK = pharmacokinetic.

- When coinciding with safety and/or PK assessments, ECGs, vital signs, and PK blood collections should be performed in said order.
- <sup>2</sup> Triplicate 12-lead ECGs will be measured at predose. Single 12-lead ECGs will be measured at all other time points.
- Urine collection intervals include 0 (predose), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 14 hours, 14 to 16 hours, 16 to 18 hours, 18 to 20 hours, 20 to 24 hours, 24 to 36 hours, 36 to 48 hours, and 48 to 60 hours.

Table 6 Safety and PK Assessments - Part 1, Period 3 (6-Hour Dose Interval)

| Procedure <sup>1</sup> | | | | | | | | | | | | | Period ( | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Predose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 6 | 6.5 | 7 | 7.5 | 8 | 8.5 | 9 | 10 | 12 | 14 | 18 | 24 | 36 | 48 | 60 |
| 12-lead ECG <sup>2</sup> | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| ECG Holter monitoring | Х | | | | | | | | | | ) | < | | | | | | | | | | | | |
| Vital signs | Χ | | | | Χ | Χ | | | Χ | | | | Χ | Χ | | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ |
| Study intervention | | Χ | | | | | | | | Х | | | | | | | | | | | | | | |
| Blood PK sample | Х | | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | Χ | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Urine PK collection <sup>3</sup> | Х | | ) | ( | | | Χ | | Χ | | ) | | | | Χ | | Χ | Χ | Χ | Х | Х | Χ | Χ | Х |

ECG = electrocardiogram; PK = pharmacokinetic.

- When coinciding with safety and/or PK assessments, ECGs, vital signs, and PK blood collections should be performed in said order.
- Triplicate 12-lead ECGs will be measured at predose. Single 12-lead ECGs will be measured at all other time points.
- Urine collection intervals include 0 (predose), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 10 hours, 10 to 12 hours, 12 to 14 hours, 14 to 18 hours, 18 to 24 hours, 24 to 36 hours, 36 to 48 hours, and 48 to 60 hours.

Table 7 Safety and PK Assessments - Part 2, Period 1

| Procedure <sup>1</sup> | | | | | | | | Treatmen<br>Time poi | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Predose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 6 | 8 | 12 | 24 | 36 | 48 |
| 12-lead ECG <sup>2</sup> | Х | Х | Х | Х | Χ | Χ | Χ | Χ | Χ | Х | Х | Х | Х | Χ | Х |
| ECG Holter monitoring | Χ | | X | | | | | | | | | | | | |
| Vital signs | Χ | | | | Х | Х | | | Х | | Х | Х | Х | Х | Х |
| Study intervention | | Х | | | | | | | | | | | | | |
| Blood PK sample | Χ | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Urine PK collection <sup>3</sup> | Χ | | ) | X | | | Χ | | Х | Х | Х | Χ | Х | Х | Х |

ECG = electrocardiogram; PK = pharmacokinetic.

Note: The number of PK samples and the PK sampling time points may be modified based on the adult PK data from Part 1.

Table 8 Safety and PK Assessments - Part 2, Period 2 (if 6-hour dose interval is selected)

| Procedure <sup>1</sup> | | | | | | | | | | | | | Period 2<br>(hours | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Predose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 6 | 6.5 | 7 | 7.5 | 8 | 8.5 | 9 | 10 | 12 | 14 | 18 | 24 | 36 | 48 | 60 |
| 12-lead ECG <sup>2</sup> | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| ECG Holter monitoring | Х | | | | | | | | | | ) | X | | | | | | | | | | | | |
| Vital signs | Χ | | | | Χ | Χ | | | Χ | | | | Χ | Χ | | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ |
| Study intervention | | Χ | | | | | | | | Х | | | | | | | | | | | | | | |
| Blood PK sample | Х | | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Χ | Х | Χ | Х | Χ | Χ | Х | Х | Χ | Χ | Х |
| Urine PK collection <sup>3</sup> | Х | | ) | ( | | | Χ | | Χ | | ) | ( | | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х |

When coinciding with safety and/or PK assessments, ECGs, vital signs, and PK blood collections should be performed in said order.

Triplicate 12-lead ECGs will be measured at predose. Single 12-lead ECGs will be measured at all other time points.

Urine collection intervals include 0 (predose), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 24 hours, 24 to 36 hours, and 36 to 48 hours.

ECG = electrocardiogram; PK = pharmacokinetic.

- When coinciding with safety and/or PK assessments, ECGs, vital signs, and PK blood collections should be performed in said order.
- <sup>2</sup> Triplicate 12-lead ECGs will be measured at predose. Single 12-lead ECGs will be measured at all other time points.
- Urine collection intervals include 0 (predose), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 10 hours, 10 to 12 hours, 12 to 14 hours, 14 to 18 hours, 18 to 24 hours, 24 to 36 hours, 36 to 48 hours, and 48 to 60 hours.

Note: The number of PK samples and the PK sampling time points may be modified based on the adult PK data from Part 1.

Table 9 Safety and PK Assessments - Part 2, Period 2 (if 12-hour dose interval is selected))

| Procedure <sup>1</sup> | | | | | | | | | | | tmen<br>e poi | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Predose | 0 | 0.5 | 1 | 1.5 | 2 | 2.5 | 3 | 4 | 6 | 8 | 12 | 12.5 | 13 | 13.5 | 14 | 14.5 | 15 | 16 | 18 | 20 | 24 | 36 | 48 | 60 |
| 12-lead ECG <sup>2</sup> | | | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| ECG Holter monitoring | Х | | | | | | | | | | Х | | | | | | | | | | | | | | |
| Vital signs | | | | | Х | Χ | | | Х | | Χ | Χ | | | Χ | Χ | | | | Χ | | Χ | Χ | Χ | Χ |
| Study intervention | | Χ | | | | | | | | | | Х | | | | | | | | | | | | | |
| Blood PK sample | Х | | Х | Χ | Х | Х | Х | Х | Χ | Χ | Χ | Х | Х | Х | Х | Χ | Х | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ |
| Urine PK collection <sup>3</sup> | Х | | Х | | | | Х | | Χ | Χ | Χ | | | X | | | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Х |

ECG = electrocardiogram; PK = pharmacokinetic.

- When coinciding with safety and/or PK assessments, ECGs, vital signs, and PK blood collections should be performed in said order.
- Triplicate 12-lead ECGs will be measured at predose. Single 12-lead ECGs will be measured at all other time points.
- Urine collection intervals include 0 (predose), 0 to 2 hours, 2 to 4 hours, 4 to 6 hours, 6 to 8 hours, 8 to 12 hours, 12 to 14 hours, 14 to 16 hours, 16 to 18 hours, 18 to 20 hours, 20 to 24 hours, 24 to 36 hours, 36 to 48 hours, and 48 to 60 hours.

Note: The number of PK samples and the PK sampling time points may be modified based on the adult PK data from Part 1.

# 10.2. Appendix 2: Study Phases and Treatment Emergent Adverse Events

#### 10.2.1. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment for the respective treatment period.

#### 10.2.1.1. Treatment States for Safety Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date/Time < Study Treatment Start Date/Time |
| On-Treatment | Study Treatment Start Date/Time ≤ Date/Time ≤ Study Treatment Stop Date/Time + 2 Days |
| Post-Treatment | Date/Time > Study Treatment Stop Date/Time +2 Days |

#### NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 10.2.1.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date/Time < Study Treatment Start Date/Time |
| On-Treatment | If AE onset date/time is on or after treatment start date/time & on or before the treatment stop date/time with 2 days lag time Study Treatment Start Date/Time ≤ AE Start Date/Time ≤ Study Treatment Stop Date/Time + 2 Days |
| Post-Treatment | If AE onset date/time is after the treatment stop date/time with 2 days lag time AE Start Date/Time > Study Treatment Stop Date/Time + 2 days |
| Onset Time<br>Since First Dose<br>(Days) | If Treatment Start Date/Time > AE Onset Date/Time = AE Onset Date - Treatment Start Date If Treatment Start Date/Time ≤ AE Onset Date/Time = AE Onset Date - Treatment Start Date +1 Missing otherwise |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF OR value is missing |

# NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

#### 10.2.1.3. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before enrollment date |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 5: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 10.2.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date/time is on or after treatment date/time &amp; on or before the treatment stop date/time with 2 days lag time.</li> <li>Study Treatment Date/Time ≤ AE Start Date/Time ≤ Study Treatment Date/Time + 2 days.</li> </ul> |

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

# 10.3.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | | |
|---|---|---|---|---|
| Study | | Treatment Group | Data Displays for Reporting | |
| Part | Code | Description | Description | Order [1] |
| 1,2 | Α | Gepotidacin single dose 1500 mg (Period 1) | Single Dose 1500 mg | 2 |
| 1,2 | В | Matching placebo (Period 1) | Placebo | 1 |
| 1 | С | Gepotidacin two 3000 mg doses given at Hour 0 and Hour 12 (Period 2) | Two 3000 mg Doses 12 h Interval | 3 |
| 1 | D | Two matching placebo doses given at Hour 0 and Hour 12 (Period 2) | Placebo | 1 |
| 1 | Е | Gepotidacin Two 3000 mg dose given at Hour 0 and Hour 6 (Period 3) | Two 3000 mg Dose 6 h Interval | 4 |
| 1 | F | Two matching placebo doses given at Hour 0 and Hour 6 (Period 3) | Placebo | 1 |
| 2 | G | Gepotidacin two 3000 mg doses<br>(Period 2; exact dosing interval to be<br>determined after Part 1 is complete) | Two 3000 mg doses 12 h Interval or 6 h Interval [2] | 3 |
| 2 | Н | Two matching placebo doses (Period 2; exact dosing interval to be determined after Part 1 is complete) | Placebo | 1 |

#### NOTES:

- 1. Order represents treatments being presented in TFL, as appropriate.
- 2. In Part 2, exact dosing interval to be determined after Part 1 is complete.

# 10.3.2. Reporting Process & Standards

# Reporting Process

#### **Software**

• The currently supported versions of SAS and WinNonlin software will be used.

# **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.1].
- For creation of ADaM datasets (ADCM/ADC1/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts described in the RAP.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures (with the exception of individual PK
    concentration-time figures, where actual relative time will be used), summaries, statistical analyses
    and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures (mean figures only for PK concentrations), summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will be considered when calculating baseline and in Table 2.9 and Table 2.10, but will not be included in any other summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

#### **Descriptive Summary Statistics**

| 2000 part o dammary ordinates | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |

#### **Graphical Displays**

Refer to IDSL Statistical Principals 7.01 to 7.13.

# 10.3.3. Reporting Standards for Pharmacokinetics

| Pharmacokinetic Concentration Data | |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (xpt format) for the non-compartmental analysis will be created according to SOP 314000(2.0). Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary Statistics, Graphical Displays and Listings | <ul> <li>Refer to IDSL PK Display Standards.</li> <li>Refer to IDSL Statistical Principle 6.06.1.</li> <li>For continuous data:</li> <li>NQs at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood.</li> <li>For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration);</li> <li>for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present)</li> <li>for summary statistics, these are set to 0 (to avoid skewing of the summary statistics)</li> <li>Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly)</li> <li>If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing).</li> <li>Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only.</li> </ul> |

| Pharmacokinetic Para | Pharmacokinetic Parameter Data |
|---|---|
| PK Parameter to be<br>Derived by<br>Programmer | The following plasma PK parameters will be derived by the Programmer: Ro Cmax, Ro AUC The following urine PK parameters will be derived by the Programmer: Ae total, Ae(t1-t2), Fe%, CLr |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | N, n, arithmetic mean, 95% CI of arithmetic mean, geometric mean, 95% CI of geometric mean, SD, SD of logged data, CV (%), and between-subject geometric coefficient of variation (CVb (%)) will be reported. $ \text{CV}_b \text{ (%)} = \sqrt{(\text{exp}(\text{SD}^2) - 1) * 100} $ (SD = SD of Ln-Transformed data) |
| Parameters Not<br>Being Ln-<br>Transformed | λz, λz lower, λz upper, and λz no. of points. |
| Parameters Not<br>Being Summarized | λz, λz lower, λz upper, and λz no. of points. |
| Listings | Include the first point, last point and number of points used in the determination of $\lambda z$ for listings. |

# 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.

#### Study Day

- Calculated as the number of days from date of study drug administration (Dose Date):
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Dose Date → Study Day = Ref Date Dose Date
  - Ref Data ≥ Dose Date → Study Day = Ref Date (Dose Date) + 1

## **Period Day**

- Calculated as the number of days from treatment date for the respective period:
  - Ref Date = Missing → Period Day = Missing
  - Ref Date < Treatment Date → Period Day = Ref Date Treatment Date
  - Ref Data ≥ Treatment Date → Period Day = Ref Date (Treatment Date) + 1

## 10.4.2. Study Population

# **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Only the year of birth will be collected. The date and month will be imputed as '30<sup>th</sup> June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

# 10.4.3. Safety

#### **Adverse Events**

# **AE'S of Special Interest**

- Cardiovascular (CV) events
- Gastrointestinal events
- Acetylcholinesterase inhibition events

#### **Adverse Events with Missing Relationship or Missing Serious Indicator**

- If the relationship to study treatment is missing for a treatment-emergent AE, it'll be considered as related to the study treatment.
- If the serious indicator "Was event serious?" is missing, the AE will be considered as SAE.
- Adverse events with missing relationship or missing serious indicator will be presented as it is in listings but will be treated as related AEs or SAEs in summary tables.
#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

#### **ECG Parameters**

#### RR Interval

- IF RR interval (millisecond [msec]) is not provided directly, then RR can be derived as:
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

- If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.
- Machine read values of RR should not be replaced with derived values.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

# 10.5. Appendix 5: Reporting Standards for Missing Data

## 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as<br/>completing all phases of the study including the follow-up visit.</li> </ul> |
| | Withdrawn participants may be replaced in the study. |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures, unless<br/>otherwise specified.</li> </ul> |
| | Early termination visits will be summarized as early termination visits. |

## 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on<br>the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the CSR. |

## 10.5.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the date of study treatment; in this case the study treatment date will be used and hence the event is considered Treatment Emergent as per Appendix 2: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is more than 2 days after the date of study treatment; in this case the study treatment date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.6. Appendix 6: Values of Potential Clinical Importance

## 10.6.1. ECG

| ECG Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| | | > 450[1] | |
| Absolute OTe Intervalia | msec | > 450[2] | ≤ 480 <sup>[2]</sup> |
| Absolute QTc Interval <sup>[3]</sup> | | > 480[2] | ≤ 500 <sup>[2]</sup> |
| | | > 500[2] | |
| Absolute PR Interval | msec | < 110[1] | > 220[1] |
| Absolute QRS Interval | msec | < 75[1] | > 110[1] |
| Change from Baseline | Change from Baseline | | |
| | msec | ≤ 30 <sup>[2]</sup> | |
| Increase from Baseline QTc[3] | msec | > 30[2] | ≤ 60 <sup>[2]</sup> |
| | msec | > 60[1] | |

#### NOTES:

- 1. Represent standard ECG values of PCI for HV studies.
- 2. Represent further subdivisions of ECG values for analysis.
- 3. Qualifying QTc events, regardless whether QTcB or QTcF, will be captured.

# 10.6.2. Vital Signs

| Vital Sign Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | millimeters of<br>mercury<br>(mmHg) | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.7. Appendix 7: Division of Microbiology and Infectious Diseases Adult Toxicity Tables for Adverse Events Assessments (2007)

## 10.7.1. Laboratory Values

Parameter values are converted to use SI units.

| HEMATOLOGY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin | 9.5 to 10.5 gm/dL | 8.0 to<br>9.4 gm/dL | 6.5 to 7.9 gm/dL | <6.5 gm/dL |
| Absolute Neutrophil<br>Count | 1000 to<br>1500 /mm <sup>3</sup> | 750 to<br>999 /mm <sup>3</sup> | 500 to 749 /mm <sup>3</sup> | <500 /mm³ |
| Platelets | 75,000 to<br>99,999 /mm <sup>3</sup> | 50,000 to<br>74,999 /mm <sup>3</sup> | 20,000 to<br>49,999 /mm <sup>3</sup> | <20,000 /mm <sup>3</sup> |
| White Blood Cells | 11,000 to<br>13,000 /mm <sup>3</sup> | 13,000 to<br>15,000 /mm <sup>3</sup> | 15,000 to<br>30,000 /mm <sup>3</sup> | >30,000 or <1000 /mm <sup>3</sup> |
| % Polymorphonuclear<br>Leukocytes + Band Cells | >80% | 90 to 95% | >95% | N/A |
| Abnormal Fibrinogen | Low: 100 to<br>200 mg/dL<br>High: 400 to<br>600 mg/dL | Low:<br><100 mg/dL<br>High:<br>>600 mg/dL | Low: <50 mg/dL<br>High: N/A | Fibrinogen associated with gross bleeding or with disseminated coagulation |
| Fibrin Split Product | 20 to 40 mcg/mL | 41 to<br>50 mcg/mL | 51 to 60 mcg/dL | >60 mcg/dL |
| Prothrombin Time (PT) | 1.01 to<br>1.25 × ULN | 1.26 to<br>1.5 × ULN | 1.51 to 3.0 × ULN | >3 × ULN |
| Activated Partial Thromboplastin (APTT) | 1.01 to<br>1.66 × ULN | 1.67 to<br>2.33 × ULN | 2.34 to 3 × ULN | >3 × ULN |
| Methemoglobin 5.0 to 9.9% | | 10.0 to 14.9% | 15.0 to 19.9% | >20% |

N/A=not applicable; ULN=upper limit of normal.

| CHEMISTRIES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 to<br>135 mEq/L | 123 to<br>129 mEq/L | 116 to 122 mEq/L | <116 mEq/L or abnormal<br>sodium with mental status<br>changes or seizures |
| Hypernatremia | 146 to<br>150 mEq/L | 151 to<br>157 mEq/L | 158 to 165 mEq/L | >165 mEq/L or abnormal sodium <i>with</i> mental status changes or seizures |
| Hypokalemia | 3.0 to 3.4 mEq/L | 2.5 to<br>2.9 mEq/L | 2.0 to 2.4 mEq/L or intensive replacement therapy of hospitalization required | <2.0 mEq/L or abnormal potassium with paresis, ileus, or life-threatening arrhythmia |
| Hyperkalemia | 5.6 to 6.0 mEq/L | 6.1 to<br>6.5 mEq/L | 6.6 to 7.0 mEq/L | >7.0 mEq/L or abnormal potassium <i>with</i> life-threatening arrhythmia |
| Hypoglycemia | 55 to 64 mg/dL | 40 to 54 mg/dL | 30 to 39 mg/dL | <30 mg/dL or abnormal<br>glucose with mental status<br>changes or coma |

| Hyperglycemia (nonfasting and no prior diabetes) | 116 to<br>160 mg/dL | 161 to<br>250 mg/dL | 251 to 500 mg/dL | >500 mg/dL or abnormal glucose with ketoacidosis or seizures |
|---|---|---|---|---|
| Hypocalcemia<br>(corrected for<br>albumin) | 8.4 to 7.8 mg/dL | 7.7 to 7.0 mg/dL | 6.9 to 6.1 mg/dL | <6.1 mg/dL or abnormal calcium with life-threatening arrhythmia or tetany |
| Hypercalcemia<br>(corrected for<br>albumin) | 10.6 to<br>11.5 mg/dL | 11.6 to<br>12.5 mg/dL | 12.6 to 13.5 mg/dL | >13.5 mg/dL or abnormal calcium <i>with</i> life-threatening arrhythmia |
| Hypomagnesemia | 1.4 to 1.2 mEq/L | 1.1 to<br>0.9 mEq/L | 0.8 to 0.6 mEq/L | <0.6 mEq/L or abnormal magnesium with life-threatening arrhythmia |
| Hypophosphatemia | 2.0 to 2.4 mg/dL | 1.5 to 1.9 mg/dL<br>or replacement<br>Rx required | 1.0 to 1.4 mg/dL intensive therapy or hospitalization required | <1.0 mg/dL or abnormal phosphate with life-threatening arrhythmia |
| Hyperbilirubinemia<br>(when accompanied<br>by any increase in<br>other liver function<br>test) | 1.1 to<br><1.25 × ULN | 1.25 to<br><1.5 × ULN | 1.5 to 1.75 × ULN | >1.75 × ULN |
| Hyperbilirubinemia<br>(when other liver<br>function tests are in<br>the normal range) | 1.1 to<br><1.5 × ULN | 1.5 to<br><2.0 × ULN | 2.0 to 3.0 × ULN | >3.0 × ULN |
| Blood urea nitrogen | 1.25 to<br>2.5 × ULN | 2.6 to 5 × ULN | 5.1 to 10 × ULN | >10 × ULN |
| Hyperuricemia (uric acid) | 7.5 to<br>10.0 mg/dL | 10.1 to<br>12.0 mg/dL | 12.1 to 15.0 mg/dL | >15.0 mg/dL |
| Creatinine | 1.1 to 1.5 × ULN | 1.6 to<br>3.0 × ULN | 3.1 to 6.0 × ULN | >6 × ULN or dialysis required |

Rx=therapy; ULN=upper limit of normal.

| ENZYMES | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Aspartate aminotransferase (AST) | 1.1 to <2.0 × ULN | 2.0 to<br><3.0 × ULN | 3.0 to<br>8.0 × ULN | >8.0 × ULN |
| Alanine aminotransferase (ALT) | 1.1 to <2.0 × ULN | 2.0 to<br><3.0 × ULN | 3.0 to<br>8.0 × ULN | >8.0 × ULN |
| Gamma to glutamyl transferase (GGT) | 1.1 to <2.0 × ULN | 2.0 to<br><3.0 × ULN | 3.0 to<br>8.0 × ULN | >8.0 × ULN |
| Alkaline Phosphatase | 1.1 to <2.0 × ULN | 2.0 to<br><3.0 × ULN | 3.0 to<br>8.0 × ULN | >8.0 × ULN |
| Amylase | 1.1 to 1.5 × ULN | 1.6 to<br>2.0 × ULN | 2.1 to<br>5.0 × ULN | >5.1 × ULN |
| Lipase | 1.1 to 1.5 × ULN | 1.6 to<br>2.0 × ULN | 2.1 to<br>5.0 × ULN | >5.1 × ULN |

ULN=upper limit of normal.

| URINALYSIS | S | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Proteinuria | 1+ or<br>200 mg to 1 gm<br>loss/day | 2 to 3+ or<br>1 to 2 gm<br>loss/day | 4+ or<br>2 to 3.5 gm loss/day | Nephrotic syndrome or >3.5 gm loss/day |
| Hematuria | Microscopic only <10 RBC/HPF | Gross, no clots >10 RBC/HPF | Gross, with or without clots, or red blood cells casts | Obstructive or required transfusion |

HPF=high powered field; RBC=red blood cells.

- 10.8. Appendix 8: Multiple Comparisons & Multiplicity
- 10.8.1. Handling of Multiple Comparisons & Multiplicity

No adjustments for multiplicity will be made.

# 10.9. Appendix 9: Abbreviations & Trade Marks

## 10.9.1. Abbreviations

| terminal-phase rate constant |
|---|
| · |
| Analysis Data Model |
| adverse event |
| adverse event of special interest |
| total unchanged drug |
| amount of drug excreted in urine in a time interval |
| area under the concentration-time curve |
| area under the concentration-time curve from time 0 (predose) extrapolated to infinite time |
| area under the concentration-time curve from time 0 (predose) to 24 hours |
| post dose administration following the first dose (plasma or urine) |
| area under the concentration-time curve from time 0 (predose) to 48 hours |
| post dose administration following the first dose (plasma or urine) |
| area under the concentration-time curve from time 0 to the time of the last |
| quantifiable concentration ((plasma or urine) |
| area under the concentration-time curve from time 0 (predose) to time tau |
| (plasma or urine) |
| body mass index |
| confidence interval |
| renal clearance of drug |
| maximum observed concentration |
| Clinical Study Report |
| Division of Microbiology and Infectious Diseases |
| electrocardiogram |
| electronic case report form |
| percentage of the given dose of drug excreted in urine |
| GlaxoSmithKline |
| informed consent form |
| Integrated Data Standards Library |
| Medical Dictionary for Regulatory Activities |
| minimum inhibitory concentration |
| · |
| milligrams |
| millimeters of mercury |
| millisecond |
| pharmacokinetic |
| corrected QT interval; the measure of time between the start of the Q wave |
| and the end of the T wave |
| corrected QT interval using the Bazett formula |
| corrected QT interval using the Fridericia formula |
| Reporting and Analysis Plan |
| serious adverse event |
| Statistical Analysis Software |
| Standard Deviation |
| schedule of activities |
| terminal phase half life |
| lag time before observation of drug concentrations |

| T <sub>max</sub> | time to reach maximum observed plasma concentration |
|------------------|-----------------------------------------------------|
| WOCBP | women of childbearing potential |

# 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| GSKDrug |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|
| MedDRA |
| WHODrug |
| WinNonlin |
| SAS |

## 10.10. Appendix 10: List of Data Displays

## 10.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables Figures | |
|------------------|----------------|-------------|
| Study Population | 1.1 to 1.10 | NA |
| Safety | 2.1 to 2.17 | 2.1 to 2.3 |
| Pharmacokinetic | 3.1 to 3.4 | 3.1 to 3.11 |
| Section | Listings | |
| ICH Listings | 1 to 48 | |
| Other Listings | 49 to 52 | |

## 10.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

# 10.10.4. Study Population Tables

| Study Po | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject D | Subject Disposition and Analysis Sets | | | | |
| 1.1 | Safety | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC [1] |
| 1.2 | Safety | ES1 | Summary of Subject Disposition | | SAC [1] |
| 1.3 | Safety | ES4 | Summary of Subject Disposition at Each Study Epoch | | SAC [1] |
| 1.4 | Screened | ES6 | Summary of Reasons for Screening Failures | | SAC [1] |
| 1.5 | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | SAC [1] |
| 1.6 | Enrolled | DV1 | Summary of Important Protocol Deviations | | SAC [1] |
| Demogra | phics and Base | eline Characteristics | | | |
| 1.7 | Safety | DM3 | Summary of Demographic Characteristics | | SAC [1] |
| 1.8 | Safety | DM5 | Summary of Race and Racial Combinations | | SAC [1] |
| 1.9 | Safety | DM11 | Summary of Age Ranges | | SAC [1] |
| 1.10 | Safety | MH4 | Summary of Current Cardiovascular and Liver Disease Related Medical Conditions | | SAC [1] |

# 10.10.5. Safety Tables

| ables | | | | |
|---|---|---|---|---|
| Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Events | | | | |
| Safety | AE5B | Summary of Adverse Events by System Organ Class and Preferred Term and Maximum Grade | | SAC [1] |
| Safety | AE5B | Summary of Drug- Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade | | SAC [1] |
| Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC [1] |
| Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC [1] |
| Safety | AE5B | Summary of Acetylcholinesterase-Inhibition Adverse Events of Special Interest by System Organ Class and Preferred Term and Maximum Grade | | SAC[1] |
| Safety | SAFE_T1 | Summary of Cumulative Grades of Acetylcholinesterase-Inhibition Adverse Events of Special Interest | | SAC [1] |
| ory Measureme | ents | | | |
| Safety | LB1 | Summary of Chemistry Change from Baseline | | SAC [1] |
| Safety | LB1 | Summary of Hematology Change from Baseline | | SAC [1] |
| Safety | UR3 | Summary of Urinalysis Dipstick Results | | SAC [1] |
| Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | | SAC [1] |
| ardiograms | | | | |
| Safety | EG1 | Summary of ECG Findings | | SAC [1] |
| | Population Events Safety | PopulationIDSL / TST ID / Example ShellEventsAE5BSafetyAE5BSafetyAE15SafetyAE16SafetyAE5BSafetyAE5BSafetySAFE_T1Ory MeasurementsSafetySafetyLB1SafetyUR3SafetyLIVER1ardiograms | Population IDSL / TST ID / Example Shell Title Events Summary of Adverse Events by System Organ Class and Preferred Term and Maximum Grade Safety AE5B Summary of Drug- Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade Safety AE15 Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) Safety AE16 Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) Safety AE5B Summary of Acetylcholinesterase-Inhibition Adverse Events of Special Interest by System Organ Class and Preferred Term and Maximum Grade Safety SAFE_T1 Summary of Cumulative Grades of Acetylcholinesterase-Inhibition Adverse Events of Special Interest of Spe | Population IDSL / TST ID / Example Shell Title Programming Notes Events Safety AE5B Summary of Adverse Events by System Organ Class and Preferred Term and Maximum Grade Safety AE5B Summary of Drug- Related Adverse Events by System Organ Class and Preferred Term and Maximum Grade Safety AE15 Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) Safety AE16 Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) Safety AE5B Summary of Acetylcholinesterase-Inhibition Adverse Events of Special Interest by System Organ Class and Preferred Term and Maximum Grade Safety SAFE_T1 Summary of Cumulative Grades of Acetylcholinesterase-Inhibition Adverse Events of Special Interest Safety LB1 Summary of Chemistry Change from Baseline Safety LB1 Summary of Hematology Change from Baseline Safety UR3 Summary of Urinalysis Dipstick Results Safety LIVER1 Summary of Liver Monitoring/Stopping Event Reporting |

| 2.12 | Safety | SAFE_T2 | Summary of Frequency of Maximum Post-Dose ECG Parameter Corrected QTc Interval | SAC [1] |
|---|---|---|---|---|
| 2.13 | Safety | SAFE_T3 | Summary of Frequency of Maximum Change from Baseline for ECG Parameter Corrected QTc Interval | SAC [1] |
| 2.14 | Safety | EG2 | Summary of Change from Baseline in ECG Values | SAC [1] |
| Vital Sign | ıs | | | |
| 2.15 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | SAC [1] |
| Cardiova | Cardiovascular Risk Factors | | | |
| 2.16 | Safety | FH1 | Summary of Family History of Cardiovascular Risk Factors | SAC [1] |
| 2.17 | Safety | SU1 | Summary of Substance Use | SAC [1] |

# 10.10.6. Safety Figures

| Safety T | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Adverse | Adverse Events | | | | |
| 2.1 | Safety | AE10 | Gastrointestinal Adverse Events of Special Interest Adverse Events | Part 1, Part 2, and combined | SAC [1] |
| 2.2 | Safety | SAFE_F1 | Plot of Distribution of Cumulative Grades of Acetylcholinesterase-<br>Inhibition Adverse Events of Special Interest | Combine Part 1 and Part 2 in one page | SAC [1] |
| 2.3 | Safety | SAFE_F2 | Plot of duration and severity of Adverse Events for Individual Participants | Part1 and Part 2 | SAC [1] |

## 10.10.7. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration Data | | | | |
| 3.1. | PK | PKCT1 | Summary of Gepotidacin Plasma Pharmacokinetic Concentration-Time Data (units) by Treatment | Paginate by study part | SAC [1] |
| 3.2. | PK | PKCT1 | Summary of Gepotidacin Urine Pharmacokinetic Concentration-<br>Time Data (units) by Treatment | Paginate by study part | SAC [1] |
| PK Deri | ived Parameters | 3 | | | |
| 3.3. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Gepotidacin Plasma Pharmacokinetic Parameters by Treatment | Parameters with units. Do not Intransform Tmax or Tlag. Paginate by study part | SAC [1] |
| 3.4. | PK<br>Parameter | PKPT4 | Summary Statistics of Derived Gepotidacin Urine Pharmacokinetic Parameters by Treatment | Parameters with units, Paginate by study part | SAC [1] |

# 10.10.8. Pharmacokinetic Figures

| Pharmac Pharmac | okinetic: Figui | res | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individua | l Concentration | n Plots | | | |
| 3.1. | PK | PKCF1P | Individual Gepotidacin Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Paginate by Study Part and<br>Treatment<br>Dashed line represents the<br>LLQ<br>Participants Overlaid | SAC [1] |
| 3.2. | PK | PKCF1P | Individual Gepotidacin Urine Concentration-Time Plots (Linear and Semi Logarithmic) | Paginate by Study Part and Treatment Dashed line represents the LLQ Participants Overlaid | SAC [1] |
| Mean / M | edian Concent | tration Plots | | · | |
| 3.3. | PK | PKCF2 | Mean (± Standard Deviation) Gepotidacin Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Treatments Overlaid; All part 1 and part 2 treatments on same page | SAC [1] |
| 3.4. | PK | PKCF2 | Mean (± Standard Deviation) Gepotidacin Urine<br>Concentration-Time Plots by Treatment (Linear and<br>Semi-Logarithmic) | Treatments Overlaid; all part 1 and part 2 treatments on the same page | SAC [1] |
| 3.5. | PK | PKCF3 | Median (Range) Gepotidacin Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | Treatments Overlaid: all part 1 and part 2 treatments on the same page | SAC [1] |

| Pharmac | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6. | PK | PKCF3 | Median (Range) Gepotidacin Urine Concentration-Time Plots by Treatment for Study Part 1 (Linear and Semi-Logarithmic) | Treatments Overlaid; all part 1 and part 2 treatments on the same page | SAC [1] |
| 3.7. | PK | PKPF1 | Scatter plot of Gepotidacin Plasma Pharmacokinetic Parameters for 1500 mg dose against Body Weight | Part 1 & Part 2, adults and adolescents shown on the same page with different symbols, with a regression line and the equation; PK Parameters: Cmax, AUC (0-∞) | SAC [1] |
| 3.8. | PK | PKPF1 | Scatter plot of Gepotidacin Body-Weight Adjusted Plasma Pharmacokinetic Parameters for 1500 mg Dose against Body Weight | If significant correlation between body weight and PK parameters, then generate an additional figure of body- weight-adjusted PK parameters versus body weight | SAC [1] |
| 3.9. | PK | PKPF1 | Scatter plot of Gepotidacin Plasma Pharmacokinetic Parameters for Two 3000 mg Doses against Body Weight | PK Parameters: Cmax and AUC(0-48); by treatment; For adults and adolescents receiving the same treatment intervals, shown them on the same page with different symbols, with a regression line and the equation; | SAC [1] |

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.10. | PK | PKPF1 | Scatter plot of Gepotidacin Body-Weight Adjusted Plasma Pharmacokinetic Parameters for Two 3000 mg Doses against Body Weight | If significant correlation<br>between body weight and PK<br>parameters, then generate an<br>additional figure of body-<br>weight-adjusted PK parameters<br>versus body weight | SAC [1] |
| 3.11. | PK | PKPF2 | BOX-Whisker plots of PK Parameters for Adults and Adolescents | PK Parameters: Cmax and AUC (0-∞) for 1500mg; Cmax and AUC (0-48) for 3000 mg two doses; 1500mg and 3000mg (various intervals) on different pages; adults and adolescents on the same page | SAC [1] |

# 10.10.9. ICH Listings

| ICH : Listi | ngs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Randomiz | ation | | | • | · |
| 1 | Randomized | CP_TA1 | Listing of Randomised and Actual Treatment | | SAC [1] |
| Subject Di | isposition | | | • | · |
| 2 | Safety | ES3 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| 3 | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation | | SAC [1] |
| 4 | Randomized | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken During the Study | | SAC [1] |
| 5 | Screened | ES7 | Listing of Reasons for Screening Failure | | SAC [1] |
| 6 | Enrolled | DV2 | Listing of Important Protocol Deviations | | SAC [1] |
| 7 | Screened | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC [1] |
| 8 | Safety | SP3 | Listing of Subjects Excluded from Any Population | | SAC [1] |
| 9 | Safety | SAFE_L1 | Listing of Subjects in Previous Clinical Trial | | SAC [1] |
| Demograp | phics | | | | · |
| 10 | Safety | DM4 | Listing of Demographic Characteristics | Include height,<br>weight and BMI | SAC [1] |
| 11 | Safety | DM10 | Listing of Race | | SAC [1] |
| Medical C | onditions and Concomit | ant Medications | | | |
| 12 | Safety | MH3 | Listing of Medical Conditions | | SAC [1] |
| 13 | Safety | CM4 | Listing of Concomitant Medications | | SAC [1] |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Exposure | , | | | | |
| 14 | Safety | SAFE_L2 | Listing of Exposure Data | | SAC [1] |
| Safety | | • | | • | |
| 15 | Safety | AE2 | Listing of Relationship Between System Organ Class and Verbatim Text | | SAC[1] |
| 16 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC [1] |
| 17 | Safety | AE9CP | Listing of All Adverse Events | | SAC [1] |
| 18 | Safety | AE9CP | Listing of Study Drug Related Adverse Events | | SAC [1] |
| 19 | Safety | AE9CPA | Listing of Serious Adverse Events | | SAC [1] |
| 20 | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study | | SAC [1] |
| 21 | Safety | SAFE_L3 | Listing of Cardiovascular Adverse Events of Special Interest | Conditional display | SAC [1] |
| 22 | Safety | SAFE_L4 | Listing of Gastrointestinal Adverse Events of Special Interest | Conditional display | SAC [1] |
| 23 | Safety | SAFE_L5 | Listing of Acetylcholinesterase-Inhibition Adverse Events of Special Interest | Conditional display,<br>Flag events with<br>onset time of 0-6hr<br>post last dose | SAC [1] |
| 24 | Safety | SAFE_L6 | Listing of Non-Gastrointestinal Acetylcholinesterase-Inhibition Adverse Events of Special Interest. | Conditional display,<br>Flag events with<br>onset time of 0-6hr<br>post last dose | SAC[1] |
| 25 | Safety | SAFE_L7 | Summary of Acetylcholinesterase-Inhibition Adverse Events of Special Interest by Treatment and by Maximum Grade of Each Participant | Conditional display | SAC[1] |

| ICH : Listin | ngs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 26 | Safety | SAFE_L8 | Listing of Liver Adverse Events | Conditional display | SAC [1] |
| 27 | Safety | SAFE_L9 | Listing of Clostridium Difficile Testing | Conditional display | SAC [1] |
| Laboratory | / Measurements | | | | |
| 28 | Safety | LB6 | Listing of Chemistry Toxicities of Grade 3 or Higher | | SAC [1] |
| 29 | Safety | LB6 | Listing of All Chemistry Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |
| 30 | Safety | LB6 | Listing of Hematology Toxicities of Grade 3 or Higher | | SAC [1] |
| 31 | Safety | LB6 | Listing of All Hematology Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |
| 32 | Safety | UR2b | Listing of Urinalysis Toxicities of Grade 3 or Higher | | SAC [1] |
| 33 | Safety | UR2b | Listing of All Urinalysis Data for Subjects with Toxicities of Grade 3 or Higher | | SAC [1] |
| ECGs | | | | | |
| 34 | Safety | EG6 | Listing of Abnormal ECG Findings | | SAC [1] |
| 35 | Safety | EG6 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC [1] |
| 36 | Safety | HM10 | Listing of Holter Abnormalities | | SAC [1] |
| 37 | Safety | EG4 | Listing of ECG Values of Potential Clinical Importance | | SAC [1] |
| 38 | Safety | EG4 | Listing of ECG Change from Baseline of Potential Clinical Importance | | SAC [1] |
| 39 | Safety | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC [1] |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Vital Signs | Vital Signs | | | | |
| 40 | Safety | VS5 | Listing of Vital Signs of Potential Clinical Importance | | SAC [1] |
| 41 | Safety | VS5 | Listing of All Vital Signs for Subjects with Potential Clinical Importance Values | | SAC [1] |
| Liver Even | Liver Events | | | | |
| 42 | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | Conditional display | SAC [1] |
| 43 | Safety | LIVER10 | Listing of Hepatobiliary Laboratory Abnormalities | Conditional display | SAC [1] |
| 44 | Safety | MH3 | Listing of Medical Conditions for Subjects with Liver Stopping Events | Conditional display | SAC [1] |
| 45 | Safety | MH3 | Listing of Plasma Concentration Data for Subjects with Liver Stopping Events | Conditional display | SAC [1] |
| 46 | Safety | SAFE_L10 | Listing of Alcohol Intake at Onset of Liver Event | Conditional display | SAC [1] |
| 47 | Safety | LIVER7 | Listing of Liver Biopsy Details | Conditional display | SAC [1] |
| 48 | Safety | LIVER8 | Listing of Liver Imaging Details | Conditional display | SAC [1] |

# 10.10.10. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharm | Pharmacokinetics | | | | |
| 49 | PK | PKCL1P | Listing of Gepotidacin Plasma Concentrations (units) by Treatment | Parts 1 and 2 combined. | SAC [1] |
| 50 | PK | PKUL1P | Listing of Gepotidacin Urine Concentrations (units) by Treatment | Parts 1 and 2 combined. | SAC [1] |
| 51 | PK<br>Parameter | PKPL1P | Listing of Gepotidacin Plasma Pharmacokinetic Parameters by Treatment | Parts 1 and 2 combined. | SAC [1] |
| 52 | PK<br>Parameter | PKPL1P | Listing of Gepotidacin Urine Pharmacokinetic Parameters by Treatment | Parts 1 and 2 combined. | SAC [1] |